CLINICAL TRIAL: NCT00200304
Title: Development and Evaluation of a SlimFast Internet Behavioral Weight Loss Program
Brief Title: Evaluation of a SlimFast Internet Behavioral Weight Loss Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 2083-00
Record Dates: First submitted 2005-09-14; First posted 2005-09-20 (Estimated); Last update posted 2013-04-24 (Estimated); Status verified 2005-09

CONDITIONS: Obesity
Keywords: Obesity; Weight loss; Internet
MeSH Terms: conditions — Obesity; Weight Loss

INTERVENTIONS:
Behavioral: Internet weight loss with SlimFast and human counseling
Behavioral: Internet weight loss with SlimFast and computer counseling
Behavioral: Internet weight loss program with SlimFast

SUMMARY:
The Internet has been used effectively in behavioral weight loss programs. Most of these programs have involved a therapist who provides email counseling. The purpose of this study was to determine whether a computer-assisted weight loss program could be developed (that would use pre-programmed computer generated messages rather than human generated messages) and whether this program would be as effective as the therapist-assisted weight loss program.

DETAILED DESCRIPTION:
Specific Aims Over 50% of Americans are overweight. These individuals are at increased risk of morbidity and mortality. Weight losses of 5-10% of body weight have been shown to lower these risks. The majority of individuals who lose weight do so on their own, without the help of formal programs. Developing ways to improve weight loss in such individuals is a major public health challenge. We believe that the Internet holds tremendous promise for reaching large numbers of overweight individuals and assisting them in their weight loss efforts. Our previous research has shown that a structured behavioral weight loss program offered via the Internet, with regular feedback from a therapist, can produce average weight losses of 9 lbs. at 6 months. The purpose of this project is to compare the weight losses achieved at 6 months using 3 different types of Internet programs, all of which are used in combination with SlimFast as the dietary component.Subject PopulationTwo hundred twenty-five overweight individuals will be recruited, aged 20-65 with a BMI of 27-40 who want to lose weight using SlimFast. Participants must be willing to attend an initial orientation and weigh-in session and follow-up weigh-in sessions and agree that they will not begin a second weight loss program within the next 12 months. Interested participants will be required to have access to a computer with Internet connection from their home or their workplace.Methods/DesignParticipants will be randomly assigned to one of three conditions: 1) SlimFast + Current SlimFast Website; 2) SlimFast + Current SlimFast Website + Computer-Generated E-mail feedback; or 3) SlimFast + Current SlimFast Website + Therapist-Assisted E-mail feedback. All 3 groups will be placed on a calorie-restricted diet (1200-1500 kcal/day) that utilizes SlimFast for 2 meals per day and a healthy evening meal. They will be encouraged to increase their exercise to 1000 kcal/week based on walking. Group 1 will receive all other input from the SlimFast website. Group 2 will receive weekly computer-generated feedback based on diet, physical activity and weight loss information. Group 3 will receive weekly e-mail messages from a trained therapist that will provide feedback based on diet, physical activity and weight loss information.Data AnalysisAll participants will be weighed at baseline, 3 months, and 6 months to document the weight changes they experience. The primary analysis will compare weight change from baseline to 6 months for the 3 conditions. An intent-to-treat analysis will be used, where dropouts are considered to have regained back to baseline weight. Secondary analyses will examine baseline predictors of weight loss and the association between use of the various Internet components and outcome.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obese

Exclusion Criteria:

* heart disease
* stroke
* cancer
* diabetes
* orthopedic problems
* pregnancy

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 225
Dates: Start 2001-01; Primary Completion 2003-01 (Actual); Study Completion 2003-01 (Actual)

PRIMARY OUTCOMES:
Weight loss at 6 months

SECONDARY OUTCOMES:
Frequency of use of the Internet website

CONTACTS AND LOCATIONS:
Overall Officials: Rena R Wing, Ph.D., Principal Investigator — The Miriam Hospital
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Result] Tate DF, Jackvony EH, Wing RR. A randomized trial comparing human e-mail counseling, computer-automated tailored counseling, and no counseling in an Internet weight loss program. Arch Intern Med. 2006 Aug 14-28;166(15):1620-5. doi: 10.1001/archinte.166.15.1620. PMID 16908795